CLINICAL TRIAL: NCT01105377
Title: Phase II Study of Azacitadine and Entinostat in Patients With Metastatic Colorectal Cancer
Brief Title: Azacitidine and Entinostat in Treating Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2010-02024; NCI-2010-02024 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000670136; MC084B (Other: Mayo Clinic); 8341 (Other: CTEP); N01CM00099 (NIH); P30CA015083 (NIH); N01CM00038 (NIH)
Record Dates: First submitted 2010-04-15; First posted 2010-04-16 (Estimated); Results first posted 2013-11-01 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Recurrent Colon Cancer; Recurrent Rectal Cancer; Stage IV Colon Cancer; Stage IV Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — entinostat; Azacitidine

ARMS (1):
- Treatment (entinostat, azacitidine) (Experimental): Patients receive azacitidine subcutaneously on days 1-5 and 8-10 and oral entinostat on days 3 and 10. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: entinostat; Drug: azacitidine; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: entinostat — Given orally
  Other Names: HDAC inhibitor SNDX-275; SNDX-275
Drug: azacitidine — Given SC
  Other Names: 5-AC; 5-azacytidine; azacytidine; Vidaza
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well giving azacitidine together with entinostat works in treating patients with metastatic colorectal cancer. Drugs used in chemotherapy, such as azacitidine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Entinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving azacitidine together with entinostat may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the preliminary efficacy via Response Evaluation Criteria In Solid Tumors (RECIST) response rate of the combination of azacitidine and entinostat in patients with metastatic colorectal cancer.

SECONDARY OBJECTIVES:

I. Explore the effects of azacitidine and entinostat on time to progression in patients with metastatic colorectal cancer.

II. To assess the toxicity for combination azacitidine and entinostat therapy.

TERTIARY OBJECTIVES:

I. Evaluate changes in promoter methylation of selected genes from DNA in circulating serum samples.

II. To determine changes in histone deacetylase activity and acetylation of H3 and H4 histones in pre- and post-treatment tumor biopsies.

III. To evaluate correlations between these molecular effects and clinical outcomes (response, time to progression).

IV. To correlate response rates by RECIST criteria versus response rates determined be EASL (change in tumor enhancement).

OUTLINE: This is a multicenter study.

Patients receive azacitidine subcutaneously on days 1-5 and 8-10 and oral entinostat on days 3 and 10. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Blood and tumor tissue samples are collected at baseline and periodically during courses 1-3 for DNA methylation, histone deacetylation activity, and acetylation of H3 and H4 histones analysis by PCR, western blot, and RT-PCR assays. Pharmacogenomic studies may also be conducted.

After completion of study therapy, patients are followed up every 3-6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic colorectal cancer
* Measurable disease
* Patient has failed ≥ 2 prior chemotherapy regimens
* Not a candidate for curative resection
* No CNS metastases within ≤ 2 years

  * Treatment for brain metastasis and whole brain disease that has remained stable for > 3 months allowed
  * Patients who have not been treated with steroid therapy may be allowed
* ECOG performance status 0-1
* Life expectancy ≥ 12 weeks
* Leukocytes ≥ 3,000/mm^3
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* Negative pregnancy test
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Sensory neuropathy ≤ grade 2 allowed
* Willing to provide tissue and blood samples
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to entinostat, azacitidine, mannitol, or other agents used in the study
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * NYHA class II-IV symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness and/or social situations that would limit compliance with study requirements
* No history of severe bleeding without thrombocytopenia
* No concurrent radiotherapy including palliative treatment
* Toxicities from prior therapy have resolved to ≤ grade 1
* More than 4 weeks since prior chemotherapy (> 6 weeks for nitrosoureas or mitomycin C)
* More than 4 weeks since prior major surgical procedure
* No prior histone deacetylase inhibitors (including valproic acid) or demethylating agents
* No concurrent investigational agents
* No concurrent combination antiretroviral therapy in HIV-positive patients
* No concurrent investigational or commercial anticancer agents or therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2010-04; Primary Completion 2012-03 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nilofer Azad, Principal Investigator — Mayo Clinic
Locations (14):
- United States (14):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of Southern California/Norris Cancer Center, Los Angeles, California
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Johns Hopkins University/Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Metro-Minnesota CCOP, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

REFERENCES:
- [Derived] Li H, Chiappinelli KB, Guzzetta AA, Easwaran H, Yen RW, Vatapalli R, Topper MJ, Luo J, Connolly RM, Azad NS, Stearns V, Pardoll DM, Davidson N, Jones PA, Slamon DJ, Baylin SB, Zahnow CA, Ahuja N. Immune regulation by low doses of the DNA methyltransferase inhibitor 5-azacitidine in common human epithelial cancers. Oncotarget. 2014 Feb 15;5(3):587-98. doi: 10.18632/oncotarget.1782. PMID 24583822

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study opened 4/12/2010, registered 24 participants (Cohort I), and suspended accrual due to toxicity on 9/10/2010. The study registered 23 participants (Cohort II) after re-opening 5/4/2011 with more restrictive eligibility criteria and closed 12/8/2011. The primary endpoint is evaluated using participants registered onto Cohort II.
Pre-assignment Details: Interim evaluation of the first 24 participants revealed more extensive disease than expected. Eligibility criteria were modified (as reflected in the Eligibility Criteria section) and registered another 23 patients (Cohort II). One patient in Cohort II cancelled prior to initiating study treatment and is not evaluable for the primary endpoint.
Groups:
- Cohort I: Treatment Prior to Eligibility Criteria Amendment: Participants 1-24 were registered according to the Eligibility Criteria for Cohort I detailed in this report. Participants received 40 mg/m^2 azacitidine subcutaneously on days 1-5 and 8-10 and 7 mg oral entinostat on days 3 and 10. Courses repeat every 28 days until disease progression or unacceptable toxicity.
- Cohort II: Treatment After Eligibility Criteria Amendment: Participants 25-47 were registered according to the eligibility requirements detailed in the Eligibility Criteria section of this report for Cohort II, which contains more restrictive criteria than Cohort I. Study treatment remained the same as Cohort I. Participants receive 40 mg/m^2 azacitidine subcutaneously on days 1-5 and 8-10 and 7 mg oral entinostat on days 3 and 10. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Cohort I | Cohort II
Started | 24 | 23
Completed | 24 | 22
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants accrued to this study are included in the description of baseline patient demographics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort I | Cohort II | Total
Number analyzed (Participants) | 24 | 23 | 47
Age, Continuous [Median (Full Range); unit: years] | 57.0 [28.0 to 75.0] | 62.6 [32.1 to 75.1] | 58.0 [28.0 to 75.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 13 | 14 | 27
Region of Enrollment [Number; unit: participants]
  United States | 24 | 23 | 47

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Tumor Response
Description: Each evaluable patient is classified as having a confirmed tumor response if they have either a complete response (CR) or partial response (PR) lasts at least 4 weeks. Tumor response is measured by using RECIST v1.1 (Response Evaluation Criteria in Solid Tumors). A CR is defined as a disappearance of all target lesions, and each target lymph node must have reduction in short axis to <1.0 cm. A PR is defined as a 30% decrease in the sum of the longest diameter for all target lesions plus the sum of the short axis of all the target lymph nodes at current evaluation, compared to pre-treatment measurements. The confirmed response rate is calculated as the number of confirmed CR+PR, divided by the total number of evaluable patients, with 95% confidence intervals estimated using the approach of Duffy and Santner.
Time Frame: At 6 month evaluation
Population: Analysis was performed "per protocol" using only Cohort II participants, except those deemed ineligible, cancelled, or in major treatment violation during cycle 1. One of the 23 Cohort II participants was excluded in the analysis due to cancelling before initiating treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort I | Cohort II
Number analyzed (Participants) | 0 | 22
percentage of participants |  | 0 [NA to NA] — A 95% Confidence Interval was not estimated due to a lack of response.

2. Secondary Outcome: Time to Progression
Description: Time to disease progression (TTP) is defined as the time from the start of treatment to the earliest of the date documenting disease progression or most recent assessment for patients having no progression. The distribution of TTP is estimated using the method of Kaplan-Meier.
Time Frame: From the start of treatment to the earliest of the date documenting disease progression, assessed up to 3 years
Population: Analysis for this endpoint was "per protocol" and two participants were excluded. One participant in Cohort I was ineligible and one participant in Cohort II refused to start their 1st cycle of study treatment (ie, cancelled). Therefore, 23 participants in Cohort I and 22 participants in Cohort II were analyzed for this secondary endpoint.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort I | Cohort II
Number analyzed (Participants) | 23 | 22
months | 1.8 [1.7 to 3.7] | 1.9 [1.8 to 2.2]

ADVERSE EVENTS:
Description: All participants receiving protocol treatment were evaluated for toxicity. 23 participants form Cohort I and 22 participants from Cohort II initiated treatment. Patients received 40 mg/m^2 azacitidine subcutaneously days 1-5 and 8-10 and 7 mg oral entinostat on days 3 and 10 in each 28 day cycle until disease progression or unacceptable toxicity.
Arm/Group | Cohort I | Cohort II
Serious Adverse Events (participants affected / at risk) | 12/24 | 5/22
Other Adverse Events (participants affected / at risk) | 24/24 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort I (N=24) | Cohort II (N=22)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (3) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (2)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 6 (18) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Erythroderma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort I (N=24) | Cohort II (N=22)
Anemia (Blood and lymphatic system disorders) | 19 (46) | 18 (35)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 7 (8) | 3 (4)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (9) | 4 (7)
Diarrhea (Gastrointestinal disorders) | 6 (7) | 2 (3)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 17 (28) | 9 (11)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 14 (19) | 5 (6)
Chills (General disorders) | 2 (3) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 19 (57) | 16 (30)
Fever (General disorders) | 2 (3) | 0 (0)
Injection site reaction (General disorders) | 4 (10) | 3 (5)
Pain (General disorders) | 0 (0) | 2 (2)
Hepatic hemorrhage (Hepatobiliary disorders) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (2)
Alkaline phosphatase increased (Investigations) | 7 (8) | 4 (6)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (2)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
CD4 lymphocytes decreased (Investigations) | 1 (2) | 0 (0)
Creatinine increased (Investigations) | 2 (4) | 0 (0)
INR increased (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 6 (11) | 3 (3)
Neutrophil count decreased (Investigations) | 1 (5) | 6 (8)
Platelet count decreased (Investigations) | 6 (8) | 7 (8)
White blood cell decreased (Investigations) | 2 (15) | 10 (16)
Anorexia (Metabolism and nutrition disorders) | 8 (11) | 7 (7)
Dehydration (Metabolism and nutrition disorders) | 2 (4) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (6) | 3 (5)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (11) | 2 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (3) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 3 (6) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 4 (9) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 3 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (3)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Uterine pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3 (4) | 2 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (12) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less